CLINICAL TRIAL: NCT05976334
Title: A Phase 1 Study to Assess Mass Balance, Pharmacokinetics, and Metabolism of [14C]Subasumstat in Patients With Advanced or Metastatic Solid Tumors
Brief Title: An Absorption, Distribution, Metabolism, Excretion (ADME) Study of [14C]Subasumstat in Adults With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-981-1004; 2023-503449-79-00 (EU CTIS Number: EU CTIS)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-981

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: [14C] Subasumstat (Experimental): Participants received a single dose of [14C] subasumstat 90 milligrams (mg), intravenous (IV) infusion on Day 1 in Part A of the study.
  Interventions: Drug: [14C] Subasumstat
- Part B: Subasumstat (Experimental): Participants received subasumstat 90 mg, IV infusion on Days 1, 4, 8, and 11 of a 21 day cycle for 3 cycles after Part A, followed by weekly maintenance dosing in Part B of the study up to maximum treatment duration of 1 year.
  Interventions: Drug: Subasumstat

INTERVENTIONS:
Drug: [14C] Subasumstat — [14C] Subasumstat IV infusion.
  Other Names: TAK-981
  Arms: Part A: [14C] Subasumstat
Drug: Subasumstat — Subasumstat IV infusion.
  Other Names: TAK-981
  Arms: Part B: Subasumstat

SUMMARY:
The main aim of this study is to assess how the human body of adults with advanced or metastatic solid tumors absorbs, distributes, metabolizes and excretes subasumstat following a single 1 hour infusion of subasumstat.

The study consists of two parts. In Part A, participants will receive a single infusion of C14 radiolabeled subasumstat. In Part B, participants will receive subasumstat treatment for up to 1 year.

DETAILED DESCRIPTION:
The drug being tested in this study is called [14C]subasumstat. [14C]Subasumstat is being tested to assess mass balance and absorption, distribution, metabolism, excretion (ADME) of people who have advanced or metastatic solid tumors.

The study will enroll approximately 10 patients. Participants will be enrolled to receive a single dose of [14C]subasumstat:

- [14C]Subasumstat 90 mg

Participants will be administered with a single dose of [14C]subasumstat 90 mg as a 1-hour intravenous (IV) infusion on Day 1 of Part A. All participants will be monitored for up to 14 days postdose. Participants will then have an option to enter Part B of the study to receive non-radiolabelled subasumstat 90 mg, IV infusion on Days 1, 4, 8, and 11 of a 21-day cycle for 3 cycles up to maximum treatment duration of 1 year.

This multi-center trial will be conducted in Hungary. The overall study duration is 12 months for Part A and 24 months for Part B.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants have histologically or cytologically confirmed advanced (locally regionally recurrent not amenable to curative therapy) or metastatic solid tumors with no standard therapeutic option with a proven clinical benefit, are intolerant or have refused them.
2. Participants have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
3. Participants demonstrate adequate organ function.
4. Participants have recovered to Grade 1 or baseline from all toxicity associated with previous therapy or have the toxicity established as sequela.

Key Exclusion Criteria:

1. Participants received treatment with radioisotopes within 5 half-lives before the first dose of the study drug.
2. Participants received radiolabelled substances, were exposed to radiation sources within 12 months of the first dose in this study, or is likely to receive radiation exposure or radioisotopes within 12 months of the first dose in this study such that participation in this study would increase their total exposure beyond the recommended safe levels.
3. Participants received extended field radiotherapy ≤4 weeks before the start of treatment.
4. Participants have uncontrolled brain metastasis. Participants with treated brain metastases are allowed provided they are radiologically stable, without evidence of progression for at least 4 weeks by repeat imaging, clinically stable, and without requirement of steroid treatment for at least 14 days before first dose of study treatment.
5. Participants had a second malignancy within the previous 3 years, except treated basal cell or localized squamous skin carcinomas, prostate cancer, cervical carcinoma in situ, resected colorectal adenomatous polyps, breast cancer in situ, or other malignancy for which the patient is not on active anticancer therapies.
6. Major surgery ≤14 days from the first dose of study drug and not recovered fully from any complications from surgery.
7. Baseline prolongation of the QT interval when corrected using Fridericia's formula (QTcF).
8. Receiving or requires the continued use of medications that are known to be strong or moderate inhibitors and inducers of cytochrome P450 (CYP) 3A4/5 and strong P-glycoprotein (Pgp) inhibitors.
9. Has active noninfectious pneumonitis or interstitial lung disease that required steroids.
10. History of allogeneic tissue or solid organ transplant.
11. Participants have active bacterial infection requiring systemic therapy <14 days before the start of treatment.
12. Participants have an active HIV or any other relevant congenital or acquired immunodeficiency.
13. Active hepatitis B, or hepatitis C infection.
14. Any of the following uncontrolled heart diseases: congestive heart failure New York Heart Association Grade III or IV, unstable angina, myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, ongoing symptomatic cardiac arrhythmias >Grade 2, pulmonary embolism or symptomatic cerebrovascular events, or any other serious cardiac condition (eg, pericardial effusion or restrictive cardiomyopathy). Chronic atrial fibrillation on stable anticoagulant therapy is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- Hungary (2):
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Pharmaceutical Research Associates Magyarorszag, Budapest

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/8c7f195d5afd4f90?idFilter=%5B%22TAK-981-1004%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 participants took part in the study at 1 investigative site in Hungary from 14 November 2023 to 16 July 2024.
Pre-assignment Details: Participants with advanced or metastatic solid tumors were enrolled in this study to receive [14C] subasumstat in Part A and subasumstat in Part B of this study.
Period: Part A
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Part B
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3
Not completed — Death | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Groups:
- Part A: [14C] Subasumstat: Participants received a single dose of [14C] subasumstat 90 mg, IV infusion on Day 1 in Part A of the study.
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percentage of Urinary Recovery
Description: Cumulative percentage of [14C]-radioactivity excreted in urine up to the last sampling interval.
Time Frame: Up to 14 days post-dose
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
percentage | 8.87 (34.5)

2. Primary Outcome: Cumulative Percentage of Fecal Recovery
Description: Cumulative percentage of [14C]-radioactivity excreted in feces up to the last sampling interval.
Time Frame: Up to 14 days post-dose
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
percentage | 75.76 (14.6)

3. Primary Outcome: Cumulative Percentage of Combined Recovery
Description: Cumulative percentage of [14C]-radioactivity excreted in urine, and feces up to the last sampling interval.
Time Frame: Up to 14 days post-dose
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
percentage | 85.27 (10.8)

4. Primary Outcome: Percentage Of Recovered Total Radioactivity (TRA) In Urine
Description: Percentage of recovered TRA in urine for each interval over the entire period of collection were reported.
Time Frame: Post-dose Day 1: 0-6 hours (hr), 6-12 hr, Day 2: 12-24 hr, Day 3: 24-48 hr, Day 4: 48-72, Day 5: 72-96 hr, Day 6: 96-120 hr, Day 7: 120-144 hr, Day 8: 144-168 hr, Day 9: 168-192 hr, Day 10: 192-216 hr, Day 11: 216-240 hr, Day 12: 240-264 hr
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug. Number analyzed is the number of participants with data available for analyses at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
mg
  Day 1- 0-6 hr | 6.11 (41.4)
  Day 1- 6-12 hr | 0.89 (36.9)
  Day 2- 12-24 hr | 0.75 (31.8)
  Day 3- 24-48 hr | 0.47 (82.6)
  Day 4- 48-72 hr | 0.18 (74.0)
  Day 5- 72-96 hr | 0.09 (52.4)
  Day 6- 96-120 hr | 0.05 (50.4)
  Day 7- 120-144 hr | 0.03 (48.5)
  Day 8- 144-168 hr | 0.03 (42.1)
  Day 9- 168-192 hr: number analyzed (Participants) | 1
  Day 9- 168-192 hr | 0.02 (NA) — Geometric coefficient of variation (%CV) was not estimable for a single participant.
  Day 10- 192-216 hr: number analyzed (Participants) | 1
  Day 10- 192-216 hr | NA (NA) — Geometric mean and %CV were not estimable for dataset containing a data point that equalled zero.
  Day 11- 216-240 hr: number analyzed (Participants) | 1
  Day 11- 216-240 hr | NA (NA) — Geometric mean and %CV were not estimable for dataset containing a data point that equalled zero.
  Day 12- 240-264 hr: number analyzed (Participants) | 1
  Day 12- 240-264 hr | NA (NA) — Geometric mean and %CV were not estimable for dataset containing a data point that equalled zero.

5. Primary Outcome: Percentage Of Recovered Total Radioactivity (TRA) In Feces
Description: Percentage of recovered TRA in feces for each interval over the entire period of collection were reported.
Time Frame: Post-dose Day 1: 0-6 hours hr, 6-12 hr, Day 2: 12-24 hr, Day 3: 24-48 hr, Day 4: 48-72 hr, Day 5: 72-96 hr, Day 6: 96-120 hr, Day 7: 120-144 hr, Day 8: 144-168 hr, Day 9: 168-192 hr, Day 10: 192-216 hr, Day 11: 216-240 hr
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Part A: [14C] Subasumstat
Number analyzed (Participants) | 3
mg
  Day 1- 0-24 hr: number analyzed (Participants) | 1
  Day 1- 0-24 hr | 0.06 (NA) — %CV was not estimable for a single participant.
  Day 3- 24-48 hr: number analyzed (Participants) | 2
  Day 3- 24-48 hr | 0.54 (131.6)
  Day 4- 48-72 hr | 63.35 (19.5)
  Day 5- 72-96 hr: number analyzed (Participants) | 1
  Day 5- 72-96 hr | 12.92 (NA) — %CV was not estimable for a single participant.
  Day 6- 96-120 hr | 4.82 (62.4)
  Day 7- 120-144 hr: number analyzed (Participants) | 2
  Day 7- 120-144 hr | 0.32 (130.0)
  Day 8- 144-168 hr | 0.26 (55.3)
  Day 9- 168-192 hr: number analyzed (Participants) | 1
  Day 9- 168-192 hr | 0.47 (NA) — %CV was not estimable for a single participant.
  Day 10- 192-216 hr: number analyzed (Participants) | 1
  Day 10- 192-216 hr | 0.16 (NA) — %CV was not estimable for a single participant.
  Day 11- 216-240 hr: number analyzed (Participants) | 1
  Day 11- 216-240 hr | 0.15 (NA) — %CV was not estimable for a single participant.

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Subasumstat and TRA in Plasma and Whole Blood
Time Frame: Pre-dose and Post-dose Day 1: 0.5 hr,1 hr,2 hr,4 hr,8 hr; Day 2: 24 hr, Day 3: 48 hr; Day 4:72 hrs; Day 5: 96 hrs; Day 6: 120 hr, Day 7: 144 hr; Day 8: 168 hr; Day 9: 192 hr,;Day 10: 216 hr; Day 11: 240 hr; Day 12: 264 hr; Day 13: 288 hr; Day 14: 312 hr
Population: The PK analysis set was planned to include participants with sufficient dosing and PK data to reliably estimate at least one PK parameter. However, due to the low number of participants and missing plasma and whole blood samples for most of them, it would not have been possible to report the data generated from these samples without compromising participant privacy. Therefore, based on the Sponsor's decision, the collected samples were not analyzed and have been disposed of.
Groups:
- All Participants: Participants received a single dose of [14C] subasumstat 90 mg, IV infusion on Day 1 in Part A of the study. Participants then received subasumstat 90 mg, IV infusion on Days 1, 4, 8, and 11 of a 21 day cycle for 3 cycles after Part A, followed by weekly maintenance dosing in Part B of the study up to maximum treatment duration of 1 year.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Subasumstat and TRA in Plasma and Whole Blood
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Subasumstat and TRA in Plasma and Whole Blood
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Terminal Disposition Phase Half-life (T1/2z) for Subasumstat and TRA in Plasma and Whole Blood as Permitted by Data
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Clearance (CL) for Subasumstat and TRA in Plasma and Whole Blood as Permitted by Data
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Volume of Distribution at Steady-state (Vss) for Subasumstat and TRA in Plasma and Whole Blood as Permitted by Data
Time Frame: as for outcome 6
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Subasumstat and TRA in Plasma and Whole Blood as Permitted by Data
Time Frame: Pre-dose and Post-dose Day 1: 0.5 hr,1 hr,2 hr 4 hr,8 hr; Day 2: 24 hr, Day 3: 48 hr; Day 4:72 hrs; Day 5: 96 hrs; Day 6: 120 hr, Day 7: 144 hr; Day 8: 168 hr; Day 9: 192 hr,;Day 10: 216 hr; Day 11: 240 hr; Day 12: 264 hr; Day 13: 288 hr; Day 14: 312 hr
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Cumulative Amount of Unchanged Subasumstat Excreted Into the Urine (Aeurine)
Description: Cumulative amount of unchanged subasumstat was determined as percentage (%) of dose of subasumstat.
Time Frame: Pre-dose and post-dose at 0-6 hours (hr) and 6-12 hr on Day 1, 12-24 hr on Day 2, 24-48 hr on Day 3, 48-72 hr on Day 4, 72-96 hr on Day 5 up to Day 14
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Mean (Standard Deviation); unit: % of dose
Arm/Group | All Participants
Number analyzed (Participants) | 3
% of dose | 8.9 (2.8)

14. Secondary Outcome: Renal Clearance (CLR) for Subasumstat in Urine
Time Frame: as for outcome 13
Population: Based on Primary Analysis results, lack of generalizability and accuracy of the urine analysis and missing data for relevant PK parameters, it would not have been possible to report the accurate data without compromising participant privacy. Therefore, based on the Sponsor's decision, the collected samples were not analyzed and have been disposed of.
Arm/Group | All Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an AE that occurred after administration of the first dose of any study drug and through 30 days after the last dose of any study drug.
Time Frame: Up to approximately 8 months
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Number analyzed (Participants) | 3 | 2
participants | 3 | 2

16. Secondary Outcome: Number of Participants With One or More Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An SAE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: Up to approximately 8 months
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Number analyzed (Participants) | 3 | 2
participants | 0 | 1

17. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram Findings
Description: Abnormal laboratory values are those outside of normal range as assessed by the investigator.
Time Frame: Up to approximately 8 months
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Number analyzed (Participants) | 3 | 2
participants | 1 | 2

18. Secondary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Laboratory findings will include serum chemistry, hematology and urinalysis. Abnormal laboratory values are those outside of normal range as assessed by the investigator.
Time Frame: Up to approximately 8 months
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: [14C] Subasumstat | Part B: Subasumstat
Number analyzed (Participants) | 3 | 2
participants
  Serum Chemistry | 3 | 2
  Hematology | 3 | 2
  Urinalysis | 0 | 1

19. Secondary Outcome: Relative Percentage of Circulatory Metabolites in Plasma
Time Frame: Pre-dose and Post-dose Day 1: 0.5 hr, 1 hr, 2 hr, 4 hr, 8 hr; Day 2: 24 hr, Day 3: 48 hr; Day 4:72 hrs; Day 5: 96 hrs; Day 6: 120 hr and Day 8: 168 hr
Population: as for outcome 6
Arm/Group | All Participants
Number analyzed (Participants) | 0

20. Secondary Outcome: Relative Percentage Excretory Metabolites in Urine
Time Frame: as for outcome 19
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Mean (Standard Deviation); unit: % of dose
Arm/Group | All Participants
Number analyzed (Participants) | 3
% of dose | 0.0 (0.0)

21. Secondary Outcome: Relative Percentage of Excretory Metabolites in Feces
Description: M1, M9 and M10 reported as categories were the names for the metabolites.
Time Frame: as for outcome 19
Population: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Measure: Mean (Standard Deviation); unit: % of dose
Arm/Group | All Participants
Number analyzed (Participants) | 3
% of dose
  Metabolite: M1 | 6.9 (1.4)
  Metabolite: M9 | 2.5 (4.3)
  Metabolite: M10 | 12.3 (2.6)

ADVERSE EVENTS:
Time Frame: Up to approximately 8 months
Description: SAS comprised of participants who had received at least 1 dose, even if incomplete, of study drug.
Groups:
- [14C] Subasumstat: Participants received a single dose of [14C] subasumstat 90 mg, IV infusion on Day 1 in Part A of the study.
- Subasumstat: Participants received subasumstat 90 mg, IV infusion on Days 1, 4, 8, and 11 of a 21 day cycle for 3 cycles after Part A, followed by weekly maintenance dosing in Part B of the study up to maximum treatment duration of 1 year.
Arm/Group | [14C] Subasumstat | Subasumstat
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [14C] Subasumstat (N=3) | Subasumstat (N=2)
General physical health deterioration (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | [14C] Subasumstat (N=3) | Subasumstat (N=2)
Aspartate aminotransferase increased (Investigations) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The enrollment for the study was halted by the sponsor for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT05976334/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT05976334/SAP_001.pdf